CLINICAL TRIAL: NCT02536001
Title: Prospective Randomized Study to Compare Anatomical, Functional and Sexual Results of Pelvic Organ Prolapse Repair With One Versus Two Vaginal Meshes While Preserving the Uterus
Brief Title: Prospective Randomized Study to Compare Results of Pelvic Organ Prolapse Repair With One Versus Two Vaginal Meshes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ziv Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0032-15-ZIV
Record Dates: First submitted 2015-07-06; First posted 2015-08-31 (Estimated); Last update posted 2015-08-31 (Estimated); Status verified 2015-05

CONDITIONS: Pelvic Organ Prolapse
Keywords: Vaginal mesh; Total vaginal length; Quality of life
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- One mesh Endofast reliant system (Other): Patients with anterior compartment stage III and uterus prolapse grade II will be treated with one mesh - Anterior Endofast reliant system (fixation of posterior arms to the sacrospinous ligament)
  Interventions: Device: One mesh Endofast reliant system
- two meshes Endofast reliant system (Other): intervention: Patients with anterior compartment stage III and uterus prolapse grade II will be treated with 2 meshes: anterior Endofast reliant system mesh to correct the anterior compartment and posterior Endofast reliant system mesh to correct the apical prolapse (fixation to the sacrospinous ligament)
  Interventions: Device: two meshes Endofast reliant system

INTERVENTIONS:
Device: One mesh Endofast reliant system — One mesh (anterior One mesh Endofast reliant system) will be used to correct both anterior and apical prolapse
  Arms: One mesh Endofast reliant system
Device: two meshes Endofast reliant system — Two meshes (anterior and posterior Endofast reliant system) will be used to correct separately the anterior compartment and the apical compartment
  Arms: two meshes Endofast reliant system

SUMMARY:
The purpose of this study is to compare anatomical differences, quality of life and sexual function and complications rate between apical support with one anterior vaginal mesh versus repair with two separate meshes.

DETAILED DESCRIPTION:
In the presence of stage 3 anterior wall prolapse (cystocele) with second stage apical prolapse (uterine or vault prolapse) there are 2 optional ways to repair with vaginal mesh: (a) to use 2 separated meshes: anterior mesh to correct the anterior compartment and posterior mesh to correct the apical prolapse to the sacrospinous ligament (SSL). (b) To correct both anterior compartment and the apical prolapse with the same mesh while using the posterior arms of the mesh to fix the apical prolapse to the SSL. Each way has its advantages and disadvantages. The first way was described at the beginning of mesh use and might be more anatomical then the second newest way. The addition of apical support to the anterior mesh might theoretically shorten the vagina. There are several recent studies describing the anatomical outcomes both for anterior compartment and apical compartment with a single mesh. Mesh-related complications, which can be also related to the amount of vaginal meshes, can potentially decrease with one mesh as compare with 2 meshes.

The aim of the study:

If the anatomical results, vaginal length and quality of life, will be with no significant differences between the two groups, the investigators will recommend to use a single mesh, in order to avoid / minimize potential complications of vaginal mesh.

If there will be no differences in complications in both groups but will be a significant difference in vaginal length and sexual function, the investigators will recommend using two meshes.

ELIGIBILITY:
Inclusion Criteria:

* At least anterior compartment prolapse stage III and uterine prolapse stage II.

Exclusion Criteria:

* Women without uterine prolapse, or with uterine prolapse < stage 2.
* Women with uterine prolapse > stage 2.
* Hysterectomy in the past.
* Women with an indication for hysterectomy.

Ages: 30 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-09; Primary Completion 2017-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Vaginal length between the arms | 2 years
  measure total vaginal length after surgery
Quality of life | 2 years
  use validated questionnaires before and after surgery
Complications rate | 2 years
  comparing complications rate between groups
Sexual function | 2 years
  use validated questionnaires before and after surgery

SECONDARY OUTCOMES:
To examine anatomical results | 2 years
  use POP-Q and compare between the groups
Success rate of uterus preservation | 2 years
  success will be define as no bulge symptoms and <stage II

CONTACTS AND LOCATIONS:
Overall Officials: Naama Marcus Braun, MD, Study Chair — Ziv Medical center, Israel